CLINICAL TRIAL: NCT06660121
Title: Treatment of Desmoid Fibromatosis With Electrochemotherapy. Prospective Observational Study
Brief Title: Electrochemotherapy for Desmoid Tumors
Acronym: ECT-DESMO
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CE AVEC: 418/2024/Oss/IOR
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Desmoid Fibromatosis
Keywords: Interventional radiology; Electrochemotherapy; Desmoid tumor
MeSH Terms: conditions — Desmoid Tumors | interventions — Electrochemotherapy; Bleomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bioptic material
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Performed electrochemotherapy: Patients diagnosed with desmoid fibromatosis unable to perform or failed other treatments who are treated with electrochemotherapy
  Interventions: Procedure: Electrochemotherapy with bleomycin

INTERVENTIONS:
Procedure: Electrochemotherapy with bleomycin — Electrochemotherapy (ECT) with bleomycin is a localized treatment approach used for managing desmoid fibromatosis, a benign but locally aggressive tumor. This technique combines electrical pulses with the administration of bleomycin, a chemotherapeutic agent, to enhance drug uptake into tumor cells. The electrical pulses create temporary pores in the cell membranes, allowing bleomycin to enter more effectively, leading to increased cytotoxicity. ECT is typically performed on patients who have not responded to conventional therapies or for whom surgery is not feasible. ECT can lead to significant tumor shrinkage and improvement in symptoms, making it a promising option in the multidisciplinary management of desmoid fibromatosis.

SUMMARY:
The goal of this observational study is to learn about the effects of Electrochemotherapy (ECT) in patients with Desmoid Fibromatosis. The main question it aims to answer is:

Is ECT effective in reducing the size of the lesion and improving patients' symptomatology?

Patients will be followed with MRI and Quality of Life questionnaires at 3, 6 and 12 months after the intervention.

DETAILED DESCRIPTION:
Desmoid fibromatoses are rare and locally aggressive, characterized histologically by monoclonal myoblasts present in abundant stromal tissue.The current therapeutic strategy has abandoned primary resection, as recurrences after resection are common and often their phenotype is more infiltrative. Nonsurgical approaches remain suboptimal. For asymptomatic disease, current guidelines suggest an initial period of active surveillance.

Other minimally invasive local treatments such as cryoablation have been shown to be effective; however, certain patients are not candidates for such treatment because of lesion location/characteristics.

An additional minimally invasive treatment with currently little evidence in the literature is arterial embolization. However, this procedure cannot be performed in the case of superficial lesions, nor in the presence of shared vasculature between the lesion and other healthy tissues or organs. In the absence of other treatments in use, electrochemotherapy treatment can be performed, which has proven effective on several other types of soft tissue and bone tumors, malignant or benign, treated at our Institute.

Electrochemotherapy is based on the principle whereby reversible electroporation causes the application of short, high-voltage electrical pulses to temporarily align water molecules on the hydrolipid layer of the cell membrane, leading to a reversible local increase in permeability by increasing the intracellular concentration of Bleomycin and its toxicity on tumor cells by a factor of up to several thousand.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Desmoid Fibromatosis and in active phase (documented growth at last follow-up)
* Patients not eligible for surgery, cryoablation, or embolization
* Signature of study-specific informed consent.

Exclusion Criteria:

* Patients with fibromatosis not in active phase, documented clinically and with imaging investigations (MRI, CT)
* Patients with documented active infection
* Previous treatment for < 30 days
* Pregnancy and lactation status
* Patients of childbearing age without contraceptive use for at least 3 months
* Presence of metal synthetic media at the site of treatment
* COPD with FiO2 < 30 mmHg
* Impaired renal function with eGFR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of desmoid fibromatosis with an indication for electrochemotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Volume reduction in cm | 1 year
  Change of the lesion evaluated with MRI, measuring the diameter of the lesion in cm.

SECONDARY OUTCOMES:
Change of pain (VAS score) | 1 year
  Clinical assessment regarding pain by Visual Analogue Scale (VAS) score (0-100 mm), in which 0 represents no pain, and 100 represents maximum pain imaginable.
Change in quality of life ( EuroQol-5D questionnaire) | 1 year
  Clinical assessment regarding quality of life by EuroQol-5D questionnaire. EQ-5D score can range from -0.594 to 1.0.
  The minimum value represents the worst possible health condition. The maximum value of 1.0 represents the best possible health condition. A value of 1.0 indicates that the patient has no problem in any of the five dimensions assessed by the questionnaire.
Feasibility of in vitro viability analysis of biopsy material | 1 year
  Evaluation of the feasibility of in vitro viability analysis of biopsy material for culturing explants and stabilizing primary cultures. Success is defined as the establishment of primary culture in 70% of samples.
  Because desmoid tumors are not aggressive, it may not be easy to maintain them in culture in vitro.
Evaluation of the role of inflammatory cytokines | 3 months
  Evaluation of the prognostic or predictive role of inflammatory cytokines detected in the blood of patients collected on the day of treatment and after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Facchini, Medicine and Surgery, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
Privacy concerns